CLINICAL TRIAL: NCT06960772
Title: Efficacy of Flow Ball Phonation in Professional Voice Users
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2025-0017
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Prevention of Voice Disorders in Professional Voice Users; Treatment of Functional Voice Disorders in Professional Voice Users
Keywords: Flow Ball; SOVTE; professional voice users; Straw Phonation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flow Ball (Experimental)
  Interventions: Behavioral: Flow Ball Intervention
- Straw Phonation (Experimental)
  Interventions: Behavioral: Straw Phonation Intervention
- Sham Intervention (Sham Comparator)
  Interventions: Behavioral: Sham Intervention

INTERVENTIONS:
Behavioral: Flow Ball Intervention — Participants receive an intensive intervention using the Flow Ball device over 3 weeks (a total of 5 hours), consisting of weekly:
  * 1 in-person guided session of 30 minutes
  * 2 guided online sessions of 15 minutes each (via teleconsult)
  * On the remaining 4 days of the week, participants perform independent training at home: 5 minutes, twice daily. This training is recorded using the app 'MyMedicoach'
  Arms: Flow Ball
Behavioral: Straw Phonation Intervention — Participants receive an intensive intervention using a straw over 3 weeks (a total of 5 hours), consisting of weekly:
  * 1 in-person guided session of 30 minutes
  * 2 guided online sessions of 15 minutes each (via teleconsult)
  * On the remaining 4 days of the week, participants perform independent training at home: 5 minutes, twice daily. This training is recorded using the app 'MyMedicoach'
  Arms: Straw Phonation
Behavioral: Sham Intervention — Participants receive an intensive intervention over 3 weeks (a total of 5 hours), consisting of weekly:
  * 1 in-person guided session of 30 minutes
  * 2 guided online sessions of 15 minutes each (via teleconsult)
  * On the remaining 4 days of the week, participants perform independent training at home: 5 minutes, twice daily. This training is recorded using the app 'MyMedicoach' The sham intervention uses breathing exercises through the Flow Ball, no phonation will be involved.
  Arms: Sham Intervention

SUMMARY:
The aim of this study is to investigate the effects of flow ball phonation on the voice of professional voice users and elite vocal performers, both with and without functional voice disorders. Given the substantial vocal demands inherent to this population and their reliance on the voice for occupational purposes, this intervention may represent a valuable approach for the prevention and/or treatment voice disorders.

DETAILED DESCRIPTION:
Background. Due to the high vocal demands, professional voice users (e.g. teachers) and elite vocal performers (e.g. singers) are risk populations for developing voice disorders. High-quality voice research in these vulnerable populations is highly needed for effective and efficient treatment and prevention of voice disorders. The flow ball (FB) is a promising innovative voice therapy device to perform semi-occluded vocal tract exercises (SOVTE) with the extra advantage of providing real-time visual feedback of the airflow. Despite this important advantage, strong efficacy studies of an FB intervention program are lacking.

Objective. To investigate the immediate-, short- and long-term effects of an SOVTE intervention with the FB on the phonation of professional voice users with (treatment) and without (prevention) voice disorders and to compare it with the 'treatment as usual' straw phonation (SP) and a sham condition, using a longitudinal randomized sham-controlled trial (RCT).

Methods. Subjects will be randomly assigned into an FB group, an SP group or a control (sham) group. They will receive a short-term intensive voice intervention of 3 weeks, combining both guided therapy/training sessions and independent practice at home. A flexible strobovideolaryngoscopy and a multidimensional voice assessment will be performed by assessors blinded to group allocation and study phase. Assessments will be performed two times before the intervention (pre 1 and pre 2), immediately after the intensive intervention (post 1) and at 3 weeks (follow-up 1) and 3 months (follow-up 2) follow-up. The sham group will use the same FB device but no phonation will be involved.

ELIGIBILITY:
OBJECTIVE 1: TREATMENT

Inclusion Criteria:

* All genders
* All ethnicities
* 18 - 60 years
* Diagnosis of a functional voice disorder
* Professional voice users

Exclusion Criteria:

* Diagnosis of an organic voice disorder
* Current participation in voice therapy
* Previous phonosurgical interventions
* Pregnancy
* Smoking
* Nasal or ear diseases
* Neurological disorders

OBJECTIVE 2: PREVENTION

Inclusion Criteria:

* All genders
* All ethnicities
* 18 - 60 years
* Professional voice users

Exclusion Criteria:

* Current or previous diagnosis of a voice disorder
* Current or previous participation in voice therapy
* Previous phonosurgical interventions
* Pregnancy
* Smoking
* Nasal or ear diseases
* Neurological disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Flexible Strobovideolaryngoscopy | baseline (before the intervention) and 3 weeks (immediately after the intervention)
  Laryngeal function determined with the Voice-Vibratory Assessment with Laryngeal Imaging (VALI) rating form (Poburka et al., 2017).
Dysphonia Severity Index (DSI) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  DSI: A higher index indicates a better voice quality. The index ranges from -5 to +5 for severely dysphonic to normal voices. A more negative index indicates a worse voice quality. Values > +5 are possible in subjects with excellent vocal capacities. A DSI = +1.6 is the threshold separating normophonic from dysphonic persons.
Acoustic Voice Quality Index (AVQI) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  A lower AVQI indicates a better voice quality. The index ranges from 0 to 10 for normal to severely dysphonic voices. An AVQI of 2.95 is the threshold separating normophonic from dysphonic persons.
Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  The CAPE-V will be used to provide an auditory-perceptual evaluation of the voice quality. This visual analogue scale will examine the voice based on the parameters grade, roughness, breathiness, asthenia, strain, instability, pitch and loudness.
Voice Handicap Index | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  VHI: A lower index indicates less impact of the voice impairment on the quality of life. The VHI ranges from 0 to 120.

SECONDARY OUTCOMES:
Maximum phonation time (MPT) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  The MPT is measured using a chronometer and the best trial out of three attempts is selected for further analysis. Participants are instructed to sustain the vowel /a:/ at their habitual pitch and loudness after a maximal inspiration. Verbal encouragement is employed to maximize phonation duration
Fundamental frequency (fo) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  To assess fo participants will produce the vowel /a:/ at their habitual pitch and loudness for three seconds, following an automatic series (counting to three).
Jitter | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  To assess the jitter participants will produce the vowel /a:/ at their habitual pitch and loudness for three seconds, following an automatic series (counting to three).
Shimmer | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  To assess the shimmer participants will produce the vowel /a:/ at their habitual pitch and loudness for three seconds, following an automatic series (counting to three).
Noise to Harmonics Ratio (NHR) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  To assess NHR participants will produce the vowel /a:/ at their habitual pitch and loudness for three seconds, following an automatic series (counting to three).
Voice Range Profile (VRP) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  The VRP indicates the vocal capabilities by examining the range of both fundamental frequency and intensity. The participants will produce the vowel /a:/ respectively at their minimum pitch, minimum intensity, maximum pitch, and maximum intensity to determine their VRP (lowest and highest fundamental frequency (Flow, Fhigh) and lowest and highest intensity (Ilow, Ihigh)).
Vocal Tract Discomfort Scale (VTDS) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  VTDS: A lower index indicates less discomfort in the vocal tract. The index ranges from 0 to 96.
Vocal Fatigue Index (VFI) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  VFI: A lower index indicates less vocal fatigue. The index ranges from 0 to 76.
Singing Voice Handicap Index 10 (SVHI-10) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  Only used with singers. The SVHI-10-NL is used assess self-perceived voice handicap among singers with singing voice difficulties. A higher index indicates a greater perceived singing voice handicap and scores of 14 or above are considered deviant. The index ranges from 0 to 40.
Evaluation of Ability to Sing Easily (EASE-NL) | baseline (twice before the intervention), 3 weeks (immediately after the intervention), 3 weeks follow-up, 3 months follow-up
  Only used with singers. The EASE-NL is a tool to assess singer's perceptions of the current status of their singing voice. It is more sensitive to detect subtle changes of the singer's voice. A higher index indicates a more deviant score. The index ranges from 0 to 60.

CONTACTS AND LOCATIONS:
Overall Officials: Evelien D'haeseleer, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No